CLINICAL TRIAL: NCT01660100
Title: Freedom From Atrial Arrhythmia in Atrial Fibrillation Patients After Permanent Pulmonary Vein Antrum Isolation With or Without Proven Left Atrial Posterior Wall Isolation
Brief Title: Outcome of Atrial Fibrillation Ablation After Permanent Pulmonary Vein Antrum Isolation With or Without Proven Left Atrial Posterior Wall Isolation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Cardiac Arrhythmia Research Foundation (Other)
Collaborators: Centro Cardiologico Monzino (Other); Catholic University of the Sacred Heart (Other); Capital Medical University (Other)
Responsible Party: Principal Investigator, Andrea Natale, Executive Medical Director, Texas Cardiac Arrhythmia Research Foundation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LIBERATION
Record Dates: First submitted 2012-08-01; First posted 2012-08-08 (Estimated); Last update posted 2017-10-19 (Actual); Status verified 2017-10

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pulmonary vein antrum isolation (PVAI) (Active Comparator): Pulmonary vein antrum isolation (PVAI)
  Interventions: Procedure: Pulmonary vein antrum isolation (PVAI)
- PVAI plus left atrial posterior wall (LAPW) isolation (Active Comparator): PVAI plus left atrial posterior wall (LAPW) isolation
  Interventions: Procedure: PVAI plus left atrial posterior wall (LAPW) isolation

INTERVENTIONS:
Procedure: Pulmonary vein antrum isolation (PVAI) — In this group, only standard PVAI will be performed during the primary procedure. Three months later, a 2nd procedure will be performed in all subjects regardless of the recurrence of atrial arrhythmias. Subjects in whom pulmonary vein antrum remains isolated will enter follow-up; however, patients who have pulmonary vein-left atrium reconnection will undergo an re-isolation. Patients who have pulmonary vein antrum re-isolation are subject to a 3rd procedure 3 months later to check the status of pulmonary vein-left atrium connection. Patients will enter follow-up for long-term outcome only after permanent PVAI is confirmed by a repeat procedure.
  Arms: Pulmonary vein antrum isolation (PVAI)
Procedure: PVAI plus left atrial posterior wall (LAPW) isolation — In this group, PVAI will be extended to the entire LAPW to achieve LAPW isolation during the primary ablation. Three months later, a 2nd procedure will be performed in all subjects regardless of the recurrence of atrial arrhythmias. Subjects in whom pulmonary vein antrum and LAPW remain isolated will enter follow-up; however, patients who have pulmonary vein antrum and/or LAPW reconnection will undergo a re-isolation. Patients who have pulmonary vein antrum and/or LAPW re-isolation are subject to a 3rd procedure three month later to check the presence of pulmonary vein antrum and/or LAPW re-connection. Patients will enter follow-up for long-term outcome only after PVAI and LAPW isolation are proven by a repeat procedure.
  Arms: PVAI plus left atrial posterior wall (LAPW) isolation

SUMMARY:
Objective: This prospective study aims to examine the outcome of atrial fibrillation (AF) ablation after permanent pulmonary vein antrum isolation or pulmonary vein antrum isolation plus left atrial posterior wall isolation is proven by a repeat procedure. The study will be conducted in patients with different types of AF: paroxysmal AF (PAF) and non-PAF (Persistent AF and Long Standing Persistent AF).

Hypothesis: In addition to permanent pulmonary vein antrum isolation, proven isolation of left atrial posterior wall is associated with more freedom from atrial arrhythmia at long-term follow-up after atrial fibrillation ablation, especially in non-PAF patients.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years
2. AF patient undergoing primary catheter ablation (first procedure)
3. Ability to give informed consent

Exclusion Criteria:

1. Previous ablation of AF
2. Bleeding disorder
3. Reversible causes of AF, such as hyperthyroidism and phaeochromocytoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2012-07; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Outcome of atrial fibrillation ablation after permanent pulmonary vein antrum isolation or proven pulmonary vein antrum plus left atrial posterior wall isolation | 12 months after pulmonary vein antrum isolation or pulmonary vein antrum plus left atrial posterior wall isolation is proven by a repeat procedure
  "Procedure success" is defined as freedom from atrial arrhythmia (atrial fibrillation, atrial flutter, atrial tachycardia) off antiarrhythmic drug during follow-up after pulmonary vein antrum isolation or pulmonary vein antrum plus left atrial posterior wall isolation is proven.
  "Procedure failure" is defined as atrial arrhythmia recurrence during follow-up after pulmonary vein antrum isolation or pulmonary vein antrum plus left atrial posterior wall isolation is proven.

SECONDARY OUTCOMES:
Long-term outcome of atrial fibrillation ablation after permanent pulmonary vein antrum isolation or proven pulmonary vein antrum plus left atrial posterior wall isolation | 24 and 36 months after pulmonary vein antrum isolation or pulmonary vein antrum plus left atrial posterior wall isolation is proven by a repeat procedure
  Patients who remain free from atrial arrhythmia (atrial fibrillation, atrial flutter, atrial tachycardia) off antiarrhythmic drug at the 12th month will be continuously followed-up every 3 months. Outcome ("Procedure success" or "Procedure failure") of atrial fibrillation ablation will be assessed at the 24th and 36th month.
Quality of life after atrial fibrillation ablation | Before atrial fibrillation ablation and 3, 6, 12 months after normal sinus rhythm is restored by successful ablation(s)

OTHER OUTCOMES:
Freedom from atrial arrhythmia (atrial fibrillation, atrial flutter, atrial tachycardia) after non-pulmonary vein trigger ablation | 6 and 12 months after re-do ablation in previously "failed" patients
  In patients who experience "procedure failure" (defined above), a re-do ablation may be performed. During the re-do procedure, in addition to re-isolation of re-connected pulmonary vein antrum and left atrial posterior wall, all non-pulmonary vein triggers will be eliminated. Then the patients will be followed-up again for atrial arrhythmia (atrial fibrillation, atrial flutter, atrial tachycardia) recurrence.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Natale, MD, Principal Investigator — Texas Cardiac Arrhythmia Insititute; Luigi Di Biase, MD, PhD, Principal Investigator — Texas Cardiac Arrhythmia Insititute; Claudio Tondo, MD, Principal Investigator — Centro Cardiologico Monzino; Rong Bai, MD, Principal Investigator — Beijing Anzhen Hospital
Locations (1):
- Texas Cardiac Arrhythmia Institute, Austin, Texas, United States

REFERENCES:
- [Derived] Bai R, Di Biase L, Mohanty P, Trivedi C, Dello Russo A, Themistoclakis S, Casella M, Santarelli P, Fassini G, Santangeli P, Mohanty S, Rossillo A, Pelargonio G, Horton R, Sanchez J, Gallinghouse J, Burkhardt JD, Ma CS, Tondo C, Natale A. Proven isolation of the pulmonary vein antrum with or without left atrial posterior wall isolation in patients with persistent atrial fibrillation. Heart Rhythm. 2016 Jan;13(1):132-40. doi: 10.1016/j.hrthm.2015.08.019. Epub 2015 Aug 13. PMID 26277862